CLINICAL TRIAL: NCT00595751
Title: Best Estimate Diagnosis Used to Evaluate EEG in Association With ADHD in a Multi-Site, Clinical Sample of Children and Adolescents
Brief Title: NeuroLex EEG-Based ADHD Assessment Aid, Pivotal Study
Acronym: NEBA
Status: Completed | Type: Observational
Sponsor: Lexicor Medical Technology, LLC (Industry)
Responsible Party: Howard Merry, President, Lexicor Medical Technology, LLC
Other Study IDs: 004-1.6
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD, Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will evaluate the effectiveness of a standardized EEG method with the intended clinical users in the intended clinical settings with the intended population (patients who would typically receive a clinician's evaluation for ADHD). Multiple sites will be examined to provide a sample of patients across numerous communities with different demographics. The goal is to evaluate if the predictive accuracy of EEG will not be inferior to that of a widely-used and extensively validated ADHD scale in the prediction of ADHD in the intended use population as evaluated by Best Estimate Diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject willing to voluntarily participate in a research study that includes EEG collection and analysis.
* Family/patient seeking comprehensive clinical evaluation for attention and/or behavior concerns.
* Male or female at least 6 years of age and who will not be over 17.99 years of age upon admission to study.
* Willing to stop any and all current psychiatric medications prior to or by entry into study.
* Subject and parent (or legal representative) of an educational level and degree of understanding sufficient to communicate suitably with the investigator, rater and study coordinator.

Exclusion Criteria:

* Previous diagnosis of mental retardation. IQ < 70 by previous records.
* History of seizure disorder or of EEG abnormalities. On anticonvulsants for seizure control.
* Metal plate or metal device in the head.
* Suicide ideation or gesture and/or homicidal ideation or gesture.
* Concomitant medications during participation in a research study. No prescription or nonprescription medications with psychoactive properties that may affect EEG (such as over-the-counter dietary supplements, pseudoephedrine, or phenylpropanolamine). No antipsychotics, no psychostimulants, no antidepressants. Washout of at least one week or longer depending on the medication and clinician's judgment. Medication used for medical reasons must be cleared by research staff with consideration of known effects on EEG.
* Known serious medical problems (cardiovascular, hematological, liver, seizure disorder, renal, or chronic respiratory problems).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study focuses on individuals who have consecutively presented to participating clinics with suspected attention and/or behavior concerns and would receive a clinician's comprehensive evaluation for ADHD. The study population includes male and female participants aged 6-17.99 years regardless of race, ethnicity, and socioeconomic origin. Because of inclusion of patients with consecutive presentation to provide a representative clinical sample, the exact numbers for sub-groups will not be controlled. The study population will include patients with comorbid conditions. The non-ADHD subgroup will include patients with other causes of attentional concerns, which may include other common psychiatric disorders, organic causes of attention problems (such as poor hearing, vision disturbances, remote head injury, substance abuse), and/or no diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
'Best Estimate Diagnosis' of ADHD applied in the intended population in settings with the intended users | At prensentation to clinic with attention or behavior problems

CONTACTS AND LOCATIONS:
Overall Officials: Humberto Quintana, MD, Study Director — LSU, HSC; Steve Snyder, Ph.D., Study Chair — Lexicor Medical Technology, LLC; Humberto Quintana, MD, Principal Investigator — LSU, HSC
Locations (10):
- United States (10):
  - Harmonex, Dothan, Alabama
  - Indian Crest Pediatrics, Westminster, Colorado
  - Medical College of Georgia, Augusta, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - LSU, HSC, New Orleans, Louisiana
  - Children's Specialized Hospital, Toms River, New Jersey
  - SUNY Upstate Medical University, Syracuse, New York
  - Rakesh Ranjan, MD & Associates, Beachwood, Ohio
  - Eminence Research, LLC, Oklahoma City, Oklahoma
  - Oklahoma University Child Study Center, Oklahoma City, Oklahoma